CLINICAL TRIAL: NCT00090025
Title: A Phase 3 Multicenter, Open Label, Randomized Study of XL119 Versus 5-Fluorouracil (5-FU) Plus Leucovorin (LV) in Subjects With Advanced Biliary Tumors Not Amenable to Conventional Surgery
Brief Title: XL119 Versus 5-Fluorouracil (5-FU) Plus Leucovorin (LV) in Subjects With Advanced Biliary Tumors
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility reasons after Independent Data Monitoring Committee interim analysis
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Helsinn Healthcare SA, Pharma Company Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XL119-001
Record Dates: First submitted 2004-08-19; First posted 2004-08-23 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Biliary Tract Cancer
Keywords: Advanced Biliary Cancer; Cholangiocarcinoma; Gall bladder tumor; Gall bladder cancer; Bile duct tumor; Tumor of biliary tree
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms; Bile Duct Neoplasms | interventions — becatecarin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- becatecarin (Experimental): becatecarin
  Interventions: Drug: becatecarin
- 5-FU Plus Leucovorin (LV) (Active Comparator): 5-Fluorouracil (5-FU) Plus Leucovorin (LV)
  Interventions: Drug: 5-Fluorouracil Plus Leucovorin

INTERVENTIONS:
Drug: becatecarin — Dose: 140 mg/m2 x day Mode of administration: i.v. via central venous catheter Duration of treatment: Days 1 through 5 of a 28 day cycle
  Other Names: XL119
  Arms: becatecarin
Drug: 5-Fluorouracil Plus Leucovorin — 5-Fluorouracil (5-FU) + Leucovorin (LV) Dose: 375 mg /m2/day + 25 mg/m2/day Mode of administration: i.v. via central venous catheter or alternative i.v. administration.Duration of treatment: Days 1 through 5 of a 28 day cycle
  Arms: 5-FU Plus Leucovorin (LV)

SUMMARY:
The main purpose of this study is to determine if XL119 is more effective than the combination of 5-fluorouracil (5FU) and leucovorin (LV) in prolonging the survival of subjects with advanced biliary tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with advanced histologically confirmed biliary cancer (gallbladder cancer or cholangiocarcinoma) that is not amenable to conventional surgical approach
* 18 years or older
* Life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) Performance Status score less than 3
* Willing and able to sign informed consent
* Sexually active men and women must use an accepted and effective method of contraception (including barrier contraception with spermicide)
* Women of child-bearing age must have a negative pregnancy test
* Laboratory criteria

Exclusion Criteria:

* Prior chemotherapy (excluding chemotherapy given as adjuvant treatment completing more than 6 months prior to entry into study)
* Unstable angina, or class III or IV New York Heart Association heart disease
* Central nervous system metastases
* Uncontrolled diabetes mellitus
* Uncontrolled seizure disorder
* Major surgery, chemotherapy, immunotherapy, or radiotherapy during the 28 days preceding the first study treatment
* Need for concomitant anticancer therapy (chemotherapy, immunotherapy, or radiation) or other investigational agents during study participation or 28 days prior to study participation
* Pregnant or breast-feeding
* A known history of human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2004-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To compare survival duration for XL119 and 5-FU/LV treated subjects | time to death

SECONDARY OUTCOMES:
To determine time to progressive disease for XL119 and 5-FU/LV treated subjects, to evaluate clinical benefit for XL119 and 5-FU/LV treated subjects, and to assess the safety profile of XL119 | time to progressive disease

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Dowlati, MD, Study Chair — Case Western Reserve University - Cleveland
Locations (59):
- United States (27):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Long Beach VA Medical Center, Long Beach, California
  - University of California, Irvine Medical Center, Orange, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Tampa General Hospital, Tampa, Florida
  - Winship Cancer Institute, Emory University Hospital, Atlanta, Georgia
  - Carle Clinic Association, Urbana, Illinois
  - Medical Consultants, PC c/o Ball Cancer Center, Muncie, Indiana
  - Oncology Associates, Cedar Rapids, Iowa
  - Louisiana Oncology Associates, Lafayette, Louisiana
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Oncology Care Center PLLC, Saint Joseph, Michigan
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Queens Hospital Center, Jamaica, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Cancer Treatment and Research Center, Bismarck, North Dakota
  - Gabrail Cancer Center, Canton, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Charleston Hematology Oncology, PA, Charleston, South Carolina
  - The Sarah Cannon Cancer Center, Nashville, Tennessee
  - Western Washington Oncology, Inc., Lacey, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Canada (5):
  - British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Centre Hospitalier Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- France (4):
  - CHU - Hospital Jean Minjoz, Besançon
  - Hospital Ambroise Pare, Boulogne-Billancourt
  - Centre Oscar Lambret, Lille
  - Institut Gustave Roussy, Villejuif
- Germany (9):
  - Charite Berlin der Humbold Universitat, Berlin
  - Heinrich-Heine-Universitat-Dusseldorf, Düsseldorf
  - Allgem. Krankenhaus St. Georg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Johannes Gutenberg, Mainz
  - Technischen Universitat Munchen, Munich
  - Klinikum Grosshadern der Ludwig Maximilians Universitaet, Munich
  - Universitätsklinikum Tübingen, Tübingen
  - Universitatsklinikum Ulm, Ulm
- Orszagos Onkologiai Intezet, Budapest, Hungary
- Italy (3):
  - Centro di Riferimento Oncologico di Aviano, Aviano
  - Ospidale Civile di Livorno, Livorno
  - Policlinico Universitario di Udine, Udine
- Centrum Onkologii - Instytut im. Marii, Warsaw, Poland
- Cancer Research Center named after N.N. Blokhin, RAMS, Moscow, Russia
- Spain (6):
  - Hospital Clinic i Provincial (Oncology Department), Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Provincial de Pontevedra, Pontevedra
  - Hospital Lozano Blesa, Zaragoza
- Leicester Royal Infirmary, Leicester, England, United Kingdom